CLINICAL TRIAL: NCT01943799
Title: A Phase 2, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of GS-4774 for the Treatment of Virally-Suppressed Subjects With Chronic Hepatitis B
Brief Title: Safety and Efficacy of GS-4774 for the Treatment of Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-330-0101
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Chronic HBV Infection
Keywords: Hepatitis B (HBV); Oral antiviral (OAV); GS-4774
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OAV Alone (Experimental): Participants will continue their prebaseline OAV regimen alone from baseline to Week 48.
  Interventions: Drug: OAV Regimen
- OAV + GS-4774 2 YU (Experimental): Participants will continue their prebaseline OAV regimen from baseline to Week 48, and will receive GS-4774 2 yeast units (YU) from baseline to Week 20.
  Interventions: Biological: GS-4774; Drug: OAV Regimen
- OAV + GS-4774 10 YU (Experimental): Participants will continue their prebaseline OAV regimen from baseline to Week 48, and will receive GS-4774 10 YU from baseline to Week 20.
  Interventions: Biological: GS-4774; Drug: OAV Regimen
- OAV + GS-4774 40 YU (Experimental): Participants will continue their prebaseline OAV regimen from baseline to Week 48, and will receive GS-4774 40 YU from baseline to Week 20.
  Interventions: Biological: GS-4774; Drug: OAV Regimen

INTERVENTIONS:
Biological: GS-4774 — Administered as a subcutaneous injection every 4 weeks for a total of 6 doses
  Arms: OAV + GS-4774 10 YU; OAV + GS-4774 2 YU; OAV + GS-4774 40 YU
Drug: OAV Regimen — Administered prior to study enrollment (tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination)

SUMMARY:
The primary objectives of this study are to evaluate the safety and efficacy of GS-4774 in adults with chronic hepatitis B (CHB) viral infection who have been virally suppressed with an oral antiviral (OAV) medication.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Currently taking an approved HBV oral antiviral medication
* Documented evidence of chronic HBV infection (eg, HBsAg positive for more than 6 months)
* Virally-suppressed (HBV DNA below the lower limit of quantification (LLOQ) for ≥ 1 year)

Key Exclusion Criteria:

* Cirrhosis
* Inadequate liver function
* Co-infection with hepatitic C virus (HCV), HIV or hepatitic D virus (HDV)
* Evidence of hepatocellular carcinoma
* Significant cardiovascular, pulmonary, or neurological disease
* Females who are pregnant or may wish to become pregnant during the study
* Received solid organ or bone marrow transplant
* Use of another investigational agents within 3 months of screening
* Current alcohol or substance abuse judged by the investigator to potentially interfere with compliance
* History of demyelinating disease (Guillain-Barre), Bell's Palsy, Crohn's disease ulcerative colitis, autoimmune disease
* Known hypersensitivity to study drug, metabolites or formulation excipients
* Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Participants under evaluation for possible malignancy are not eligible.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2015-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (17):
- United States (16):
  - Dumont-UCLA Liver Transplant Center, Los Angeles, California
  - Huntington Medical Research Institutes, Pasadena, California
  - Kaiser Permanente, Sacramento, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Miami, Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital and Health System, Detroit, Michigan
  - St.Louis University, St Louis, Missouri
  - Medical Pro-care, Flushing, New York
  - North Shore LIJ Health System, Manhasset, New York
  - Bon Secours St. Mary's Hospital of Richmond, Newport News, Virginia
- Auckland Clinical Studies, Grafton, New Zealand

REFERENCES:
- [Derived] Lok AS, Pan CQ, Han SH, Trinh HN, Fessel WJ, Rodell T, Massetto B, Lin L, Gaggar A, Subramanian GM, McHutchison JG, Ferrari C, Lee H, Gordon SC, Gane EJ. Randomized phase II study of GS-4774 as a therapeutic vaccine in virally suppressed patients with chronic hepatitis B. J Hepatol. 2016 Sep;65(3):509-16. doi: 10.1016/j.jhep.2016.05.016. Epub 2016 May 19. PMID 27210427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States and New Zealand. The first participant was screened on 13 September 2013. The last study visit occurred on 03 March 2015.
Pre-assignment Details: 213 participants were screened.
Groups:
- OAV Alone (Group A): Participants continued to receive their prebaseline oral antiviral (OAV) regimen alone from baseline to Week 48. Prebaseline OAV regimen may have included the following: tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination.
- OAV + GS-4774 2 YU (Group B): Participants continued to receive their prebaseline OAV regimen from baseline to Week 48 and received GS-4774 2 yeast units (YU) administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Prebaseline OAV regimen may have included the following: tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination.
- OAV + GS-4774 10 YU (Group C): Participants continued to receive their prebaseline OAV regimen from baseline to Week 48 and received GS-4774 10 YU administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Prebaseline OAV regimen may have included the following: tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination.
- OAV + GS-4774 40 YU (Group D): Participants continued to receive their prebaseline OAV regimen from baseline to Week 48 and received GS-4774 40 YU administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Prebaseline OAV regimen may have included the following: tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination.
Period: Overall Study
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Started | 27 | 50 | 51 (1 participant was randomized to OAV + GS-4774 2 YU but received OAV + GS-4774 10 YU.) | 50
Completed | 22 | 47 | 49 | 50
Not Completed | 5 | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who had a Group A Baseline visit or received at least 1 dose of GS-4774 for Group B, C, and D. For each participant, the average of non-missing doses were calculated and participants were assigned based on the average: Group A = 0 YU, Group B = > 0 and ≤ 6 YU, Group C = > 6 YU and ≤ 25 YU, or Group D = > 25 YU.
Groups:
- OAV Alone (Group A): Participants continued to receive their prebaseline OAV regimen alone from baseline to Week 48. Prebaseline OAV regimen may have included the following: tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination.
- OAV + GS-4774 2 YU (Group B): Participants continued to receive their prebaseline OAV regimen from baseline to Week 48 and received GS-4774 2 YU administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Prebaseline OAV regimen may have included the following: tenofovir disoproxil fumarate, entecavir, adefovir, lamivudine, or telbivudine either as single agents or in combination.
- Total: Total of all reporting groups
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D) | Total
Number analyzed (Participants) | 27 | 50 | 51 | 50 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10.9) | 50 (9.0) | 47 (10.0) | 47 (11.1) | 47 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 14 | 19 | 56
  Male | 20 | 34 | 37 | 31 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 27 | 48 | 50 | 49 | 174
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 21 | 40 | 41 | 34 | 136
  White | 5 | 6 | 3 | 7 | 21
  Other | 1 | 3 | 4 | 2 | 10
  Black or African American | 0 | 1 | 2 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: 1 participant from the United States was randomized to OAV + GS-4774 2 YU but received OAV + GS-4774 10 YU.
  Participants
    New Zealand | 4 | 6 | 2 | 7 | 19
    United States | 23 | 44 | 49 | 43 | 159
Hepatitis B Surface Antigen (HBsAg) (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 2.5 (1.46) | 3.1 (0.72) | 3.0 (1.02) | 3.0 (0.86) | 2.9 (0.99)
HBsAg Level [Count of Participants; unit: Participants]
  ≤ 1000 IU/mL | 13 | 18 | 21 | 21 | 73
  > 1000 IU/mL | 14 | 32 | 30 | 29 | 105
Hepatitis B Envelope Antigen (HBeAg) Status [Count of Participants; unit: Participants]
  Positive | 7 | 13 | 12 | 12 | 44
  Negative | 20 | 37 | 39 | 38 | 134

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HBsAg at Week 24
Description: The change from baseline to Week 24 in HBsAg was analyzed using a mixed effect model for repeated measures (MMRM). The model included included treatment, HBsAg baseline level (≤ 1000 IU/mL or > 1000 IU/mL), HBeAg baseline status (positive or negative), visit, and treatment-by-visit interaction as fixed effects and visit as a repeated measure.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set (participants who were randomized and had a Baseline/Day 1 visit for Treatment Group A or have received at least 1 dose of GS-4774 for Treatment Group B, C, and D) with available data were analyzed. Participants were analyzed according to the randomized treatment assignment.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 21 | 47 | 48 | 49
log10 IU/mL | -0.019 [-0.070 to 0.031] | -0.020 [-0.055 to 0.014] | -0.026 [-0.060 to 0.008] | -0.048 [-0.082 to -0.014]
Statistical Analysis 1: Comparison: OAV Alone (Group A) vs OAV + GS-4774 2 YU (Group B); Each null hypothesis was tested against the 2-sided alternative that the mean change from baseline in serum HBsAg (log10 IU/mL) titers in the respective GS-4774 group was not equal to that of the OAV group. Estimated least squares means (LSM) of treatment effects and estimated differences in treatment effects between GS-4774 treatment groups and the OAV group at Week 24 were calculated with 95% confidence intervals (CIs) and unadjusted p-values; Test type: Superiority; p = 0.976, MMRM; LS Mean Difference = -0.001, 95% CI 2-sided [-0.061 to 0.059]
Statistical Analysis 2: Comparison: OAV Alone (Group A) vs OAV + GS-4774 10 YU (Group C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.828, MMRM; LS Mean Difference = -0.007, 95% CI 2-sided [-0.067 to 0.053]
Statistical Analysis 3: Comparison: OAV Alone (Group A) vs OAV + GS-4774 40 YU (Group D); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.343, MMRM; LS Mean Difference = -0.029, 95% CI 2-sided [-0.089 to 0.031]

2. Secondary Outcome: Change From Baseline in HBsAg at Week 12
Description: The change from baseline to Week 12 in HBsAg was analyzed using a MMRM. The model included included treatment, HBsAg baseline level (≤ 1000 IU/mL or > 1000 IU/mL), HBeAg baseline status (positive or negative), visit, and treatment-by-visit interaction as fixed effects and visit as a repeated measure.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 21 | 48 | 49 | 49
log10 IU/mL | -0.004 [-0.041 to 0.033] | -0.016 [-0.041 to 0.010] | -0.017 [-0.043 to 0.008] | -0.028 [-0.054 to -0.003]

3. Secondary Outcome: Change From Baseline in HBsAg at Week 48
Description: The change from baseline to Week 48 in HBsAg was analyzed using a MMRM. The model included included treatment, HBsAg baseline level (≤ 1000 IU/mL or > 1000 IU/mL), HBeAg baseline status (positive or negative), visit, and treatment-by-visit interaction as fixed effects and visit as a repeated measure.
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 20 | 48 | 48 | 49
log10 IU/mL | -0.043 [-0.179 to 0.094] | -0.055 [-0.148 to 0.038] | -0.051 [-0.143 to 0.041] | -0.166 [-0.257 to -0.075]

4. Secondary Outcome: Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 24
Description: HBsAg loss was defined as HBsAg level decreasing from >0.066 IU/mL at baseline to ≤ 0.066 IU/mL at any postbaseline visit. HBsAb seroconversion was defined as HBsAb level increasing from < 12 mIU/mL at baseline to ≥ 12 mIU/mL at any postbaseline visit.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with HBsAg Level above 0.066 IU/mL at Baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 25 | 50 | 50 | 50
percentage of participants
  HBsAg Loss | 0 | 0 | 0 | 0
  HBsAg Loss and Seroconversion | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 48
Description: as for outcome 4
Time Frame: Week 48
Population: Participants in the Full Analysis Set with HBsAg Level above 0.066 IU/mL at Baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 25 | 50 | 50 | 50
percentage of participants
  HBsAg Loss | 0 | 0 | 0 | 0
  HBsAg Loss and Seroconversion | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With HBeAg Loss and HBeAg Seroconversion by Week 24
Description: HBeAg loss was defined as a qualitative HBeAg result changing from positive at baseline to negative at any postbaseline visit. HBeAb seroconversion was defined as a qualitative HBeAb result changing from negative at baseline to positive at any postbaseline visit.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with positive HBeAg at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 7 | 13 | 12 | 12
percentage of participants
  HBeAg Loss | 0 | 0 | 25.0 | 0
  HBeAg Loss and Seroconversion | 0 | 0 | 25.0 | 0

7. Secondary Outcome: Percentage of Participants With HBeAg Loss and HBeAg Seroconversion by Week 48
Description: as for outcome 6
Time Frame: Week 48
Population: Participants in the Full Analysis Set with positive HBeAg at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 7 | 13 | 12 | 12
percentage of participants
  HBeAg Loss | 0 | 7.7 | 33.3 | 0
  HBeAg Loss and Seroconversion | 0 | 7.7 | 25.0 | 0

8. Secondary Outcome: Percentage of Participants With a 1-log Decline in HBsAg by Weeks 12, 24, and 48
Description: HBsAg 1-log decline was defined as ≥ 1 decline from baseline in log10 IU/mL serum HBsAg at any postbaseline visit within the targeted time window.
Time Frame: Baseline; Weeks 12, 24, and 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
Number analyzed (Participants) | 27 | 51 | 50 | 50
percentage of participants
  ≥ 1 log10 IU/mL Decline at Week 12 | 0 | 0 | 0 | 0
  ≥ 1 log10 IU/mL Decline at Week 24 | 0 | 0 | 0 | 0
  ≥ 1 log10 IU/mL Decline at Week 48 | 0 | 0 | 0 | 2.0

ADVERSE EVENTS:
Time Frame: First dose date up to Week 20 plus 28 days
Description: The Safety Analysis Set included participants who have had a Baseline/Day 1 visit for Group A or have received at least one dose of GS-4774 for Group B, C, and D. For each participant, the average of non-missing doses of GS-4774 were calculated. The participant was assigned to Group A if the average was 0, or Group B if the average was greater than 0 and no more than 6 YU, or Group C if the average was greater than 6 YU and no more than 25 YU, or Group D if the average was greater than 25 YU.
Arm/Group | OAV Alone (Group A) | OAV + GS-4774 2 YU (Group B) | OAV + GS-4774 10 YU (Group C) | OAV + GS-4774 40 YU (Group D)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/50 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/50 | 1/51 | 0/50
Other Adverse Events (participants affected / at risk) | 7/27 | 39/50 | 47/51 | 46/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAV Alone (Group A) (N=27) | OAV + GS-4774 2 YU (Group B) (N=50) | OAV + GS-4774 10 YU (Group C) (N=51) | OAV + GS-4774 40 YU (Group D) (N=50)
Colonic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OAV Alone (Group A) (N=27) | OAV + GS-4774 2 YU (Group B) (N=50) | OAV + GS-4774 10 YU (Group C) (N=51) | OAV + GS-4774 40 YU (Group D) (N=50)
Nausea (Gastrointestinal disorders) | 0 | 3 | 4 | 6
Chills (General disorders) | 0 | 2 | 5 | 7
Fatigue (General disorders) | 0 | 8 | 13 | 13
Injection site erythema (General disorders) | 0 | 18 | 29 | 36
Injection site induration (General disorders) | 0 | 18 | 21 | 23
Injection site pain (General disorders) | 0 | 19 | 34 | 39
Injection site pruritus (General disorders) | 0 | 13 | 16 | 26
Injection site swelling (General disorders) | 0 | 12 | 17 | 25
Pyrexia (General disorders) | 0 | 1 | 0 | 4
Influenza (Infections and infestations) | 2 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 5 | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 7 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 2 | 2
Headache (Nervous system disorders) | 1 | 9 | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 6 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 2
Hypertension (Vascular disorders) | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years